CLINICAL TRIAL: NCT03628469
Title: Proactive Health Support - a Randomized Controlled Trial of Telephone-based Self-management Support
Brief Title: Proactive Health Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Ulla Toft, Senior Researcher, Principal Investigator, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SJ-677
Record Dates: First submitted 2018-08-01; First posted 2018-08-14 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Patients at Risk of Hospital Admission

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 1:1 randomization stratified for risk of hospital admission and region
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive Health Support (Experimental): The purpose of the intervention is to enhance patients' self-management strategies and thereby enable patients to cope with illness at home and prevent the development of those conditions, that are sensitive to preventive efforts.The intervention includes active listening, coaching and counselling and elements from case management such as assessing the need for healthcare services. Emphasis is on supporting and empowering the patient to make the necessary contacts to healthcare professionals.
  Interventions: Behavioral: Proactive Health Support
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Proactive Health Support — Active listening, coaching and counselling
  Arms: Proactive Health Support

SUMMARY:
Proactive Health Support is a randomized controlled trial of telephone-based self-management support. The primary aim of the intervention is to reduce hospital admissions and improve quality of life in patients with a high risk of hospital admission.

DETAILED DESCRIPTION:
Participants are identified through an algorithm, that assigns each patient with a risk score of 0-100%. Patients with the highest risk in each of the five regions of Denmark are invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a hospital contact within the last year caused by ≥ 1 of the following diagnoses: heart diseases (DI110, DI130, DI132, DI50), connective tissue diseases (DD86, DM05, DM06, DM08, DM09, DM30, DM31, DM32, DM33, DM34, DM35, DM36), pulmonary diseases (DJ40, DJ41, DJ42, DJ43, DJ44, DJ45, DJ46, DJ47, DJ60, DJ61, , DJ62, DJ63, DJ64, DJ65, DJ66, DJ67, DJ684, DJ701, DJ703, DJ841, DJ842, DJ843, DJ848, DJ849, DJ920, DJ961, DJ982, DJ983) or diabetes (DE10, DE11, DE14) Or
* Persons ≥ 18 years and ≥ three unplanned hospital admissions in the last six months Or
* Persons ≥ 65 years with a preventable hospital admission (predefined diagnoses: dehydration, constipation, lower respiratory tract infections, urinary tract infections, gastroenteritis, fractures, nutrition deficiency anemia, social causes and pressure ulcers) or a readmission (within 30 days)

Exclusion Criteria:

* Selected psychiatric diagnoses: substance abuse disorder (DF1), schizophrenia (DF2) or dementia (DF00, DF01, DF02, DF03, DF051)
* Metastatic cancer (DC77, DC78, DC79, DC80)
* Assisted living Facility
* Documented terminal illness or life expectancy < one year
* Assessment of dementia
* Major surgery planned within 6 months
* Hearing impairment
* Not speaking Danish
* Cognitive impairment
* Substance abuse, that impairs adherence
* No telephone
* Receiving similar trial intervention
* Other (including intervention not suitable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5454 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Hospital admissions | 6 months
Quality of life | 6 months
  Questionnaire SF 36 - Mental Health Composite Score (Norm-based T-score of 45-55 is considered normal)

SECONDARY OUTCOMES:
Patient education | 3, 6 and 12 months
  Questionnaire Hei-Q - all 8 subscales (health-directed activities, positive and active engagement in life, emotional distress, self-monitoring and insight, constructive attitudes and approaches, skill and technique acquisition, social integration and support, health service navigation, range 1-4)
Outpatient consultations | 3, 6 and 12 months
Use of primary healthcare | 3, 6 and 12 months
Use of prescription medication | 3, 6 and 12 months
Survival | 1 year
Quality of life | 3, 6 and 12 months
  Questionnaire SF36: All eight subscales (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, mental health and health transition, range 0-100. Furthermore, norm-based T-scores are reported, 45-55 is considered normal) and two composite scores (mental and physical health, norm-based T-score of 45-55 is considered normal)
Incremental cost effectiveness ratio by comparison of costs with quality adjusted life years | 3, 6 and 12 months
Regional differences in resource use and costs | 3, 6 and 12 months
Resource use in primary care and rehabilitation | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Toft, PhD, Principal Investigator — Frederiksberg University Hospital
Locations (1):
- Center for Clinical Research and Prevention, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benthien KS, Rasmussen K, Nielsen CP, Hjarnaa L, Rasmussen MK, Kidholm K, Nielsen BK, Nissen NK, Fredens M, Winther S, Gronkjaer M, Toft U. Proactive health support (PaHS) - telephone-based self-management support for persons at risk of hospital admission: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2020 Jun;93:106004. doi: 10.1016/j.cct.2020.106004. Epub 2020 Apr 19. PMID 32320846